CLINICAL TRIAL: NCT07392736
Title: A Phase I/IIa Clinical Trial of AL8326 Tablets Combined With Toripalimab in the Treatment of Advanced Recurrent or Metastatic Solid Tumors
Brief Title: A Phase I/IIa Study of AL8326 Combined With Toripalimab in the Treatment of Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advenchen Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AL8326-CN-006
Record Dates: First submitted 2025-09-28; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AL8326 plus toripalimab (Experimental): Phase 1: Cohort 1 will initiate with AL8326 +Toripalimab 240mg multiple dose (28-Day cycles) After three subjects have completed the first cycle of therapy without a DLT, additional cohorts may be enrolled sequentially. After the first cohort has completed one full cycle of therapy without a DLT, further cohorts will be enrolled sequentially, following the same 28-day cycle regimen.
  Phase 2a: Each subject will receive AL8326 +Toripalimab 240mg of this study for continuous 28-Day/21-Day cycles of therapy. AL8326 is orally administered daily at the RP2D found in Phase 1.
  Interventions: Drug: AL8326 tablets; Drug: Toripalimab

INTERVENTIONS:
Drug: AL8326 tablets — Tablet: 10mg/tablet; administered orally once daily
  Other Names: AL8326
Drug: Toripalimab — 240mg Injection solution：21-Day cycles

SUMMARY:
This trial is an open, non-randomized, phase I/IIa clinical trial, which will evaluate the preliminary effectiveness and safety of AL8326 tablets in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria

1. Subjects must be able to understand and voluntarily sign a written informed consent form prior to the initiation of any study-related procedures.
2. Age ≥ 18 years.
3. Subjects with histologically confirmed advanced recurrent or metastatic solid tumors who meet one of the following conditions:

   1. Failure of standard therapy (disease progression after treatment or intolerance to treatment toxicity);
   2. no effective treatment available.
   3. Toripalimab monotherapy as a second-line or later standard treatment.
4. Must have at least one measurable lesion as defined by RECIST 1.1.
5. Prior cytotoxic chemotherapy must have been completed at least 4 weeks before enrollment, and any toxicities must have recovered to ≤ Grade 1 (except alopecia).
6. Life expectancy of ≥ 12 weeks at the time of enrollment.
7. ECOG performance status of 0 or 1.
8. Adequate organ function:

   1. Bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L (1500/mm³); Platelets ≥ 100 × 10⁹/L; Hemoglobin ≥ 9.0 g/dL.
   2. Renal function: Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or calculated creatinine clearance (Cockcroft-Gault formula) ≥ 60 mL/min.
   3. Hepatic function: Total bilirubin ≤ 1.5 × ULN (≤ 3.0 × ULN for subjects with Gilbert's syndrome); AST and ALT ≤ 2.5 × ULN in subjects without liver metastases, or ≤ 5 × ULN in subjects with liver metastases.
   4. Coagulation function: International normalized ratio (INR) ≤ 1.5; Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
9. Left ventricular ejection fraction (LVEF) > 50% during screening.
10. Systolic blood pressure < 140 mmHg and diastolic blood pressure < 90 mmHg (without medication or controlled with a single agent).
11. Females: Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment and must agree to use medically acceptable methods of contraception during the treatment period and for 3 months after the last dose; The patient must be non-lactating; Postmenopausal women (≥ 12 months of amenorrhea without other causes) or surgically sterilized (oophorectomy and/or hysterectomy) are not considered of childbearing potential. Their partners must use medically acceptable contraception during the treatment period and for 3 months after the last dose. Males: Surgically sterile or must agree to use medically acceptable contraception during the treatment period and for 3 months after the last dose; Their partners must use medically acceptable contraception during the same period.
12. Ability and willingness to comply with the study protocol for the duration of the study and with follow-up procedures.

Exclusion Criteria

1. Received systemic cytotoxic therapy or investigational therapy within 28 days prior to initiation of study treatment, or non-cytotoxic, non-investigational therapy (e.g., radiotherapy, hormone therapy, targeted therapy, immunotherapy) within 14 days prior to initiation of study treatment.
2. Major surgery (defined as requiring general anesthesia within 28 days before initiation of study treatment, or minor surgery requiring general anesthesia within 7 days before initiation of study treatment).
3. Pregnant or lactating women.
4. History of prior or concurrent second primary malignancy that, in the opinion of the investigator or sponsor, may interfere with the assessment of safety or efficacy of the study treatment.
5. Subjects with active or untreated central nervous system (CNS) metastases; Subjects with stable brain metastases may be enrolled if they meet the following criteria: a) No radiological evidence of progression for ≥ 4 weeks after completion of treatment; b) Completion of treatment ≥ 28 days before the first dose of study drug; c) No requirement for systemic corticosteroids (>10 mg/day prednisone or equivalent) within ≤ 14 days prior to the first dose of study drug.
6. Active, known, or suspected autoimmune disease or interstitial lung disease.
7. Requirement for systemic therapy with corticosteroids or other immunosuppressive drugs within 14 days prior to initiation of study treatment.
8. Peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with risk of perforation; History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to initiation of study treatment.
9. Untreated deep vein thrombosis (DVT) within the past 6 months. Subjects with DVT treated with therapeutic anticoagulants (excluding therapeutic warfarin) for at least 14 days prior to initiation of study treatment are allowed.
10. Uncontrolled infection.
11. New York Heart Association (NYHA) Grade III or greater congestive heart failure.
12. History of any of the following cardiac conditions within 6 months prior to initiation of study treatment:

    1. Cardiac angioplasty or stenting;
    2. Myocardial infarction;
    3. Unstable angina;
    4. Cerebrovascular accident.
13. Presence of any unhealed wound, fracture, or ulcer, or symptomatic peripheral vascular disease.
14. Evidence of hemorrhagic diathesis, coagulation disorder, or clinically significant bleeding (e.g., severe hematuria, gastrointestinal bleeding, hemoptysis) within 6 months prior to initiation of study treatment.
15. QTcF ≥470 msec on screening ECG per Fridericia's formula.
16. Urinalysis showing urine protein ≥ ++ and 24-hour urine protein quantification > 1.0 g within 28 days prior to initiation of study treatment.
17. Positive hepatitis B surface antigen (HBsAg) with HBV-DNA above the lower limit of detection of the local laboratory; Positive hepatitis C antibody (anti-HCV) with HCV-RNA above the lower limit of detection of the local laboratory; Positive syphilis antibody; Positive human immunodeficiency virus (HIV) antibody test.
18. History of organ transplantation.
19. Clinical conditions affecting the intake or absorption of AL8326 (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, malabsorption disorders, gastrectomy or small bowel resection).
20. Use of prohibited concomitant medications within 14 days prior to initiation of study treatment.
21. Receipt of red blood cell or platelet transfusion within 14 days prior to initiation of study treatment.
22. Known allergy, hypersensitivity, or intolerance to protein therapies, or history of any severe drug allergy (e.g., anaphylaxis, hepatotoxicity, immune-mediated thrombocytopenia or anemia).
23. Any severe and/or unstable pre-existing medical, psychiatric, or other condition that may jeopardize subject safety, obtaining informed consent, compliance with study procedures, or achievement of study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2029-11-07 (Estimated); Study Completion 2029-11-07 (Estimated)

PRIMARY OUTCOMES:
The first part (Phase I): Phase II recommended dose (RP2D) | At the end of Cycle 1 (each cycle is 28 days)
  Determine the Recommended Phase 2 Dose (RP2D) via evaluation of dose limiting toxicity (DLT) events.
The second part (Phase IIa):Objective remission rate (ORR) | Every 2/3/4 cycles,up to 24 month（each cycle is 21 days）
  (ORR):The proportion of subjects achieving complete remission (CR) and partial remission (PR) with optimal efficacy according to RECIST 1.1.

SECONDARY OUTCOMES:
The first part (Phase I): Objective remission rate (ORR) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  (ORR):The proportion of subjects achieving complete remission (CR) and partial remission (PR) .
The first part (Phase I): Duration of remission (DOR) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  (DOR):Description: The time between the start of the first assessment of the tumor as CR or PR and The first assessment of disease progression (PD) or death from any cause.
The first part (Phase I): Disease Control Rate (DCR) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  (DCR): The proportion of subjects achieving complete remission (CR), partial remission (PR) and stable disease (SD).
The first part (Phase I): Duration of Disease Control (DDC) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  (DDC): The time from the first assessment of the tumor as CR, PR, or SD to the first assessment of disease progression (PD) or death from any cause.
The first part (Phase I): Progression Free Survival (PFS) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  (PFS): The period of time between the start of the subject's first dose of medication and the first observation of disease progression (based on imaging) or the occurrence of death due to any cause.
The first part (Phase I): Overall Survival (OS) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  (OS): Defined as the time between the date of first dose and death from any cause. Subjects who are alive as of the date of analysis will use and the date they last achieved survival as the cutoff time.
The second part (Phase IIa): Duration of remission (DOR) | Every 2/3/4 cycles,up to 24 month（each cycle is 21 days）
  (DOR):Description: The time between the start of the first assessment of the tumor as CR or PR and The first assessment of disease progression (PD) or death from any cause.
The second part (Phase IIa): Disease Control Rate (DCR) | Every 2/3/4 cycles,up to 24 month（each cycle is 21 days）
  (DCR): The proportion of subjects achieving complete remission (CR), partial remission (PR) and stable disease (SD).
The second part (Phase IIa): Duration of Disease Control (DDC) | Every 2/3/4 cycles,up to 24 month（each cycle is 21 days）
  (DDC): The time from the first assessment of the tumor as CR, PR, or SD to the first assessment of disease progression (PD) or death from any cause.
The second part (Phase IIa): Progression Free Survival (PFS) | Every 2/3/4 cycles,up to 24 month（each cycle is 21 days）
  (PFS): The period of time between the start of the subject's first dose of medication and the first observation of disease progression (based on imaging) or the occurrence of death due to any cause.
The second part (Phase IIa): Overall Survival (OS) | Every 2/3/4 cycles,up to 24 month（each cycle is 21 days）
  (OS): Defined as the time between the date of first dose and death from any cause. Subjects who are alive as of the date of analysis will use and the date they last achieved survival as the cutoff time.

CONTACTS AND LOCATIONS:
Overall Officials: Jing wang, Principal Investigator — Hunan Cancer Hospital; LingYIng Wu, Principal Investigator — The Cancer Hospital of the Chinese Academy of Medical Sciences
Locations (15):
- China (15):
  - National GCP Center for Anticancer Drugs,The Independent Ethics Committee, Beijing, Beijing Municipality
  - The Cancer Hospital of the Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Hunan, Changsha
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - The First Affiliated Hospital of Guilin Medical Universty, Guilin, Guangxi
  - Liuzhou Workers' Hospital, Liuchow, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - SIR RUN RUN SHAW Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang